CLINICAL TRIAL: NCT03257176
Title: Stepping Stones and Creating Futures Intervention Pilot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of KwaZulu (Other)
Collaborators: Medical Research Council, South Africa (Other); Project Empower (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSS/0789/011
Record Dates: First submitted 2017-08-07; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Physical Violence; Sexual Violence; Livelihoods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stepping Stones and Creating Futures (Experimental): Receive the 21 session intervention
  Interventions: Behavioral: Stepping Stones and Creating Futures

INTERVENTIONS:
Behavioral: Stepping Stones and Creating Futures — 21 session intervention, comprising of 10 Stepping Stones sessions focused on gender, relationships and communication. 11 Creating Futures sessions focused on livelihoods.

SUMMARY:
This is a shortened interrupted time series pilot evaluation over a twelve month period to evaluate whether the combined Stepping Stones and Creating Futures intervention can reduce men's perpetration of IPV and women's experience of IPV, strengthen livelihoods and reduce gender inequality.

ELIGIBILITY:
Inclusion Criteria:

* Over 18
* Mentally competent
* Able to communicate in English, Zulu, or Xhosa
* Normally resident in the informal settlement

Exclusion Criteria:

* Over 30
* Unable to do informed consent

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 232 (Actual)
Dates: Start 2012-05-02 (Actual); Primary Completion 2013-07-30 (Actual); Study Completion 2013-07-30 (Actual)

PRIMARY OUTCOMES:
Past three month physical IPV perpetration (men) and experience (women) | 12 months post baseline
  Physical intimate partner violence is assessed using five items based on the WHO VAW scale, asking about perpetration (men) and experience (women) of these five behaviourally specific actions in the past three months. A positive response to any of the five items leads to a person being classified as perpetrating (men) and experiencing (women) physical IPV in the past three months.
Past three month sexual IPV perpetration (men) and experience (women) | 12 months post baseline
  Sexual intimate partner violence is assessed using three items based on the WHO VAW scale for sexual IPV. Questions are asked for the past three month perpetration (men) and experience (women). A positive response to any item leads to a person being classified as perpetrating (men) and experiencing (women) in the past three months.
Earnings in past month | 12 months post baseline
  A single item question asks "Considering all the money you earned from jobs or selling things (excluding grants), how much did you earn last month?" Responses are in Rands and a continuous scale.

SECONDARY OUTCOMES:
Work stress | 12 months post baseline
  4 items ask about work stress because of a lack of work. Responses are on a likert scale.
Feelings about work shame | 12 months post baseline
  4 items ask about shame because of type and lack of work. Responses are on a likert scale.
Gender attitudes | 12 months post baseline
  Modified gender equitable men's scale assess participant's gender attitudes.
Controlling behaviours | 12 months post baseline
  Controlling behaviours are assessed using a modified Sexual Relationship Power (SRP) scale. Men's control of female sexual partner's and women's experience of controlling behaviours from a male partner.
Condom use at last sex | 12 months post baseline
  Single item asking about condom use at last sex
Hunger in the past month | 12 months post baseline
  Single item assesses hunger in the past month

CONTACTS AND LOCATIONS:
Locations (1):
- Gender and Health Research Unit, South African Medical Research Council, Durban, KwaZulu-Natal, South Africa

REFERENCES:
- [Background] Gibbs A, Willan S, Jama-Shai N, Washington L, Jewkes R. 'Eh! I felt I was sabotaged!': facilitators' understandings of success in a participatory HIV and IPV prevention intervention in urban South Africa. Health Educ Res. 2015 Dec;30(6):985-95. doi: 10.1093/her/cyv059. PMID 26590246
- [Result] Jewkes R, Gibbs A, Jama-Shai N, Willan S, Misselhorn A, Mushinga M, Washington L, Mbatha N, Skiweyiya Y. Stepping Stones and Creating Futures intervention: shortened interrupted time series evaluation of a behavioural and structural health promotion and violence prevention intervention for young people in informal settlements in Durban, South Africa. BMC Public Health. 2014 Dec 29;14:1325. doi: 10.1186/1471-2458-14-1325. PMID 25544716